CLINICAL TRIAL: NCT02964806
Title: Development and Clinical Validation of Ketogen-based Therapeutic Diet for Pancreaticobiliary Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2016-0799
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Ketogen-based Therapeutic Diet; Pancreaticobiliary Cancer
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ordinary Diet (Other): Ordinary Diet
  Interventions: Dietary Supplement: Ordinary Diet
- Modified Atkin's Diet (Other): Modified Atkin's Diet
  Interventions: Dietary Supplement: Modified Atkin's Diet
- Ketogenic Diet (Other): Ketogenic Diet
  Interventions: Dietary Supplement: Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Ordinary Diet
  Arms: Ordinary Diet
Dietary Supplement: Modified Atkin's Diet
  Arms: Modified Atkin's Diet
Dietary Supplement: Ketogenic Diet
  Arms: Ketogenic Diet

SUMMARY:
Decreased bowel function and loss of appetite in patients who underwent pancreaticobiliary surgery contribute impaired nutritional status in postoperative period. It can also affect perioperative and oncologic outcomes negatively. Therefore it is important to improve nutritional status in postoperative period by supply tailor-made optimal diets. The investigators have developed customized postoperative diets for pancreaticobiliary cancer patients. The investigators expect that customized diets for pancreaticobiliary patients will increase the food intake rate and contribute a improvement of perioperative outcomes and even oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age more than 19)
* Pancreaticobiliary cancer patient who is scheduled pancreaticoduodenectomy or distal pancreatectomy
* Pancreatic cancer / Duodenal cancer / Distal bile duct cancer / Ampulla of Vater cancer

Exclusion Criteria:

* Patient who denied clinical trial
* Diabetes Mellitus(DM) patient with DM complication
* Hyperlipidemia patient with vascular co-morbidity
* Impaired renal function or renal failure (GFP<90%)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Food Intake Rate(%) for postoperative diet | 3 days after the diet
  Diet Intake Rate(%) will be examined by dietary satisfaction questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No